CLINICAL TRIAL: NCT05437042
Title: Does Medial Calcaneal Wedge Improve Static Balance and Load Distribution in Young Adults With Pronated Foot?
Brief Title: Effect of Medial Wedge on Static Balance in Pronated Feet
Status: Completed | Type: Observational
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Izgi Guven, Research Assistant, Pamukkale University
Other Study IDs: HU/PAU/GUVEN-001
Record Dates: First submitted 2022-06-23; First posted 2022-06-29 (Actual); Last update posted 2022-07-06 (Actual); Status verified 2022-07

CONDITIONS: Foot; Deformity, Valgus, Congenital; Foot; Deformity, Valgus (Acquired); Foot Deformities; Flatfoot
Keywords: Foot Orthoses; Postural Balance; Subtalar Joint
MeSH Terms: conditions — Congenital Abnormalities; Genu Valgum; Foot Deformities; Flatfoot

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Individuals with pronated foot
  Interventions: Other: Medial calcaneal wedge

INTERVENTIONS:
Other: Medial calcaneal wedge — Immediate effect of medial calcaneal wedge for static balance and weight distribution

SUMMARY:
The use of heel wedges is often recommended as a clinical routine in individuals with foot pronation. However, there is a lack of information for examining the immediate effect of supports used to restore foot biomechanics on balance. The aim of our study is to examine the immediate effect of calcaneal support in the frontal plane on static balance in individuals with increased pronated foot. In this study, the fore-hind foot load distribution in static bipedal stance will be examined in healthy young adults. Then, static balance measurements will be made on one leg with and without support (medial heel wedge). For the evaluation of static balance on one leg, x-y mean, ellipse surface, A-P index measurements and romberg test will be used. In addition, the pain of individuals will be questioned and their foot postures will be evaluated. Healthy young adult individuals with a subtalar angle of 5 degrees and above in the weighted position will be included in the evaluations. Evaluations of the participants are planned to take approximately 15 minutes.

DETAILED DESCRIPTION:
In a normal foot, the subtalar joint is pronated from heel strike to sole contact, which makes the midtarsal joint and forefoot flexible. Between sole contact and toe lift, the subtalar joint becomes supinated and the foot turns into a rigid lever (1,2). Hindfoot overpronation can be defined as pronation of the subtalar joint during gait phases in which supination is normal. It can cause problems such as abnormal pronation in the foot, increased flexibility, deterioration in load distribution, hallux valgus and heel spurs, and postural disorders involving the leg, knee, hip and spine (3). In addition, the increase in rear foot pronation negatively affects the physical performance of individuals such as jumping and running (4). Commonly used conservative methods to prevent pronation in the subtalar joint include exercises to support the medial arch, strengthen muscles and ligaments, electrical stimulation, insoles, wedges, and applications such as flexible and inflexible taping techniques (1,5).

Medial wedge is a method frequently preferred by physiotherapists in terms of ease of use among the methods used in the routine. It is thought that the contact of the medial longitudinal arch support of the insole with the foot prevents the increase in pronation of the foot and reduces the load on the arch structures. The medial longitudinal arch support transfers the load on the heel region to the midfoot and the decrease in maximum pressure in the 2nd and 3rd metatarsal regions is explained by the insoles turning the foot towards supination. It is stated that excessive pronation of the hindfoot and the secondary deformities it may cause can be prevented by the use of simple supports applied under the foot.

The foot is located at the most distal point and acts as the support base for this kinematic chain. For this reason, the smallest dynamic change in the foot affects the balance of the whole body (6). Balance is the ability to keep the body's center of gravity within the acceptable limits of the support surface during activities such as sitting, standing or walking, and it is a complex process that includes versatile sensory, motor and biomechanical components (7).

It is known that foot deformities in seniors negatively affect balance and cause falls (8). Along with the changes in the gravity line in neurological diseases, problems are seen in maintaining the balance starting from the sitting level and in situations that require a change in movement. Conditions such as loss of balance or inability to maintain body position in athletes may prevent the athlete from performing the expected performance, as well as cause injuries (9). Balance improvement has an important place in every field of physiotherapy. Improving balance, increasing function in the athlete, improving performance; To ensure the continuity of mobility in neuromuscular diseases and neurological problems, to increase the quality of life; in healthy individuals, it is important to prevent injuries. In this study, the immediate effect of the medial heel wedge on static balance and weight distribution in individuals with pronated foot was investigated.

ELIGIBILITY:
Inclusion Criteria:

* Standing subtalar angle of 5° or more
* Foot Posture Index score of 6 or more
* Right lower limb dominance
* Agreeing to participate in the study voluntarily

Exclusion Criteria:

* Having a neurological or orthopedic problem
* Having any surgery on the lower extremity
* Having a foot-ankle complex Visual Analog Scale (VAS) pain score above 6.4

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Young adults who has pronated foot
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
Immediate effect of medial heel wedge on static balance | Day 1

SECONDARY OUTCOMES:
Immediate effect of medial heel wedge on load distribution | Day 1

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University, Faculty of Physical Therapy and Rehabilitation, Ankara, Sıhhiye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Leung AK, Mak AF, Evans JH. Biomedical gait evaluation of the immediate effect of orthotic treatment for flexible flat foot. Prosthet Orthot Int. 1998 Apr;22(1):25-34. doi: 10.3109/03093649809164454. PMID 9604273
- [Background] McPoil TG, Hunt GC. Evaluation and management of foot and ankle disorders: present problems and future directions. J Orthop Sports Phys Ther. 1995 Jun;21(6):381-8. doi: 10.2519/jospt.1995.21.6.381. PMID 7655482
- [Background] Valmassy RL. clinical biomechanics of the lower extermities. Mosby, Missouri. 1996;12:143-5.
- [Background] Kararti C, Bilgin S, Buyukturan O, Buyukturan B. Arka Ayaktaki Pronasyon Artisinin Fiziksel Performans Uzerine Etkisi. Hacettepe University Faculty of Health Sciences Journal. 2018;5(1):1-0.
- [Background] Hadley A, Griffiths S, Griffiths L, Vicenzino B. Antipronation taping and temporary orthoses. Effects on tibial rotation position after exercise. J Am Podiatr Med Assoc. 1999 Mar;89(3):118-23. doi: 10.7547/87507315-89-3-118. PMID 10095333
- [Background] Al Abdulwahab SS, Kachanathu SJ. The effect of various degrees of foot posture on standing balance in a healthy adult population. Somatosens Mot Res. 2015;32(3):172-6. doi: 10.3109/08990220.2015.1029608. Epub 2015 Sep 7. PMID 26400632
- [Background] Winter DA. Human balance and posture control during standing and walking. Gait & posture. 1995 Dec 1;3(4):193-214.
- [Background] Whitney KA. Foot deformities, biomechanical and pathomechanical changes associated with aging including orthotic considerations, Part II. Clin Podiatr Med Surg. 2003 Jul;20(3):511-26, x. doi: 10.1016/S0891-8422(03)00046-6. PMID 12952051
- [Background] Borklu T, Dolu N. Sporcularda Isitsel Uyarilma Potansiyellerindeki Hemisferik Farkliliklar. Sağlık Bilimleri Dergisi (Journal of Health Sciences). 2010;19(2):108-18.